CLINICAL TRIAL: NCT06431087
Title: Effect of a Mindfulnes Program "Healthy Under Stress" on Stress and Stress-associated Parameters: A Prospective Intervention Study
Brief Title: Effect of a Mindfulnes Program "Healthy Under Stress" on Stress: A Prospective Intervention Study
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S00822-NIM
Record Dates: First submitted 2024-05-16; First posted 2024-05-28 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-05

CONDITIONS: Subjective Stress
Keywords: Mindfulness; Healthy Lifestyle
MeSH Terms: conditions — Subjective Stress

STUDY DESIGN:
Intervention Model Description: Single-Center, an Arm, prospective intervention study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulnes "Healthy Under Stress" Stress Management Program (Experimental): Participants will have two-hour sessions for 8 weeks.
  Interventions: Other: Mindfulness course

INTERVENTIONS:
Other: Mindfulness course — Online or in presence Information on Mindfulness, healthy diet and exercise.

SUMMARY:
Stress describes a state of worry and mental tension that results from an imbalance between demands and coping strategies, as well as the disruption of physiological homeostasis. It represents an important ability to adapt to environmental factors, and chronically has negative psychological and physical consequences. The mind-body medical program "Healthy in Stress" according to Esch aims to strengthen the individual's ability to deal with stress through comprehensive training. The main target parameter is stress reduction, measured using the Perceived Stress Scale (PSS).

DETAILED DESCRIPTION:
After baseline (t0), all participant will receive the following intervention:

The intervention lasts eight weeks, with a two-hour session held once a week. The selected topics include nutrition, mindfulness, exercise, relaxation techniques, dealing with stressors, effective communication and the promotion of a supportive social network.

t1 (at the end of the program).

t2 (3 months after t0).

ELIGIBILITY:
Inclusion Criteria:

* Employees, patients and family members of the Robert-Bosch-Krankenhaus (RBK) and Bosch Health Campus of all specialties.
* Informed consent.

Exclusion Criteria:

* Physical or mental condition which, in the opinion of the investigator does not allow the patient to participate in the study.
* Participation in other clinical studies with behavioral, psychological or complementary medical interventions.
* Insufficient knowledge of the German language.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-07-08 (Estimated); Primary Completion 2027-08-30 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale | After 8 Weeks (end of intervention)
  The Perceived Stress Scale (PSS-10) is a scale records patients' subjective stress in the last month in four subscales: worries, anxiety, happiness and needs). Ten items are rating on a five-point scale (1 = never, 5 = very often).

SECONDARY OUTCOMES:
Perceived Stress Scale | Follow-up 3 Moths after the intervention
  The Perceived Stress Scale (PSS-10) is a scale records patients' subjective stress in the last month in four subscales: worries, anxiety, happiness and needs). Ten items are rating on a five-point scale (1 = never, 5 = very often).
Hospital Anxiety and Depression Scale | After 8 Weeks (end of intervention)
  Hospital Anxiety and Depression Scale (HADS) is a self-report questionnaire on the severity of symptoms of anxiety and depressive disorders in the past week. The 14 items (seven on depression and seven on anxiety) are rated on a four-point scale. Each question is scored between zero (no impairment) and four (severe impairment).
Hospital Anxiety and Depression Scale | Follow-up 3 Moths after the intervention
  Hospital Anxiety and Depression Scale (HADS) is a self-report questionnaire on the severity of symptoms of anxiety and depressive disorders in the past week. The 14 items (seven on depression and seven on anxiety) are rated on a four-point scale. Each question is scored between zero (no impairment) and four (severe impairment).
Quality of life Questionnaire | After 8 Weeks (end of intervention)
  Quality of life Questionnaire (SF-36) includes one multi-item scale that assesses eight health concepts: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). Scores range from 0 - 100 (Lower scores = more disability, higher scores = less disability).
Quality of life Questionnaire | Follow-up 3 Moths after the intervention
  Quality of life Questionnaire (SF-36) includes one multi-item scale that assesses eight health concepts: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH). Scores range from 0 - 100 (Lower scores = more disability, higher scores = less disability).
International Physical Activity Questionnaire | After 8 Weeks (end of intervention)
  The International Physical Activity Questionnaire (IPAQ) records physical activity over the past seven days using 8 questions. The duration of activities of moderate and high exertion as well as the duration of sitting are asked, and the result is indicated using the metabolic equivalent (MET).
International Physical Activity Questionnaire | Follow-up 3 Moths after the intervention
  The International Physical Activity Questionnaire (IPAQ) records physical activity over the past seven days using 8 questions. The duration of activities of moderate and high exertion as well as the duration of sitting are asked, and the result is indicated using the metabolic equivalent (MET).
Mediterranean Diet Adhrence Screener | After 8 Weeks (end of intervention)
  The Mediterranean Diet Adhrence Screener (MEDAS) is a questionnaire to assess adherence to the Mediterranean diet (DM). It consists of 14 items on eating habits, each of which is rated with one or zero points. The higher the score, the better the adherence to the MD.
Mediterranean Diet Adhrence Screener | Follow-up 3 Moths after the intervention
  The Mediterranean Diet Adhrence Screener (MEDAS) is a questionnaire to assess adherence to the Mediterranean diet (DM). It consists of 14 items on eating habits, each of which is rated with one or zero points. The higher the score, the better the adherence to the MD.
Mindful Attention and Awareness Scale | After 8 Weeks (end of intervention)
  The Mindful Attention and Awareness Scale (MAAS) is a questionnaire of 15 items on a six-point scale (1 = almost always, 6 = almost never) to measure the frequency of actual experiences.
Mindful Attention and Awareness Scale | Follow-up 3 Moths after the intervention
  The Mindful Attention and Awareness Scale (MAAS) is a questionnaire of 15 items on a six-point scale (1 = almost always, 6 = almost never) to measure the frequency of actual experiences.
Safety evaluation | After 8 Weeks (end of intervention)
  In order to evaluate the safety of the intervention, unforeseen events are documented. For this purpose participants are explicitly asked about the occurrence of these.

CONTACTS AND LOCATIONS:
Overall Officials: Marcela Winkler, Dr, Study Director — Robert Bosch Gesellschaft für Medizinische Forschung mbH (RBMF)
Locations (1):
- Robert-Bosch-Krankenhaus, Stuttgart, Baden Würtenberg, Germany